CLINICAL TRIAL: NCT06790303
Title: A Phase II, Randomized, Open-label Platform Trial Utilizing a Master Protocol to Study Novel Regimens Versus Standard of Care Treatment in NSCLC Participants
Brief Title: Platform Trial of Novel Regimens Versus Standard of Care (SoC) in Participants With Non-small Cell Lung Cancer (NSCLC) - Sub-study 2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to low enrolment of participants
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205801-002; 2018-001316-29 (EudraCT Number)
Record Dates: First submitted 2025-01-22; First posted 2025-01-24 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Neoplasms
Keywords: NSCLC; Feladilimab; Iplimumab
MeSH Terms: conditions — Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Feladilimab plus Ipilimumab (Experimental)
  Interventions: Drug: Feladilimab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Feladilimab — Feladilimab will be administered.
Drug: Ipilimumab — Ipilimumab will be administered

SUMMARY:
This study is a sub-study of the master protocol 205801 (NCT03739710). This sub study will assess the clinical activity of novel regimen (Feladilimab plus Ipilimumab) in participants with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of giving signed informed consent/assent.
* Male or female, aged 18 years or older at the time consent is obtained. Participants in Korea must be age 19 years or older at the time consent is obtained.
* Participants with histologically or cytologically confirmed diagnosis of NSCLC (squamous or non-squamous) and
* Participants capable of giving signed informed consent/assent.
* Male or female, aged 18 years or older at the time consent is obtained. Participants in Korea must be age 19 years or older at the time consent is obtained.
* Participants with histologically or cytologically confirmed diagnosis of NSCLC (squamous or non-squamous) and

  1. Documented disease progression based on radiographic imaging, during or after a maximum of 2 lines of systemic treatment for locally/regionally advanced recurrent, Stage IIIb/Stage IIIc/Stage IV or metastatic disease. Two components of treatment must have been received in the same line or as separate lines of therapy: i) No more than or less than 1 line of platinum-containing chemotherapy regimen, and ii) No more than or less than 1 line of Programmed cell death ligand 1 (PD[L]1) monoclonal antibody (mAb) containing regimen.
  2. Participants with known V-Raf Murine Sarcoma Viral Oncogene Homolog B (BRAF) molecular alterations must have had disease progression after receiving the locally available SoC treatment for the molecular alteration.
  3. Participants who received prior anti-PD(L)1 therapy must fulfill the following requirements: i) Have achieved a CR, PR or SD and subsequently had disease progression (per RECIST 1.1 criteria) either on or after completing PD(L)1 therapy ii) Have not progressed or recurred within the first 12 weeks of PD(L)1 therapy, either clinically or per RECIST 1.1 criteria
* Measurable disease, presenting with at least 1 measurable lesion per RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
* A tumor tissue sample obtained at any time from the initial diagnosis of NSCLC to time of study entry is mandatory. Although a fresh tumor tissue sample obtained during screening is preferred, archival tumor specimen is acceptable.
* Adequate organ function as defined in the protocol.
* A male participant must agree to use a highly effective contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions apply:

  i) Not a woman of childbearing potential (WOCBP) or ii) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
* Life expectancy of at least 12 weeks.

Exclusion Criteria:

* Participants who received prior treatment with the following therapies (calculation is based on date of last therapy to date of first dose of study treatment):

  1. Docetaxel at any time.
  2. Any of the investigational agents being tested in the current study.
  3. Systemic approved or investigational anticancer therapy within 30 days or 5 half-lives of the drug, whichever is shorter. At least 14 days must have elapsed between the last dose of prior anticancer agent and the first dose of study drug is administered.
  4. Prior radiation therapy: permissible if at least one non-irradiated measurable lesion is available for assessment per RECIST version 1.1 or if a solitary measurable lesion was irradiated, objective progression is documented. A wash out of at least 2 weeks before start of study drug for radiation of any intended use is required.
* Received greater than (>)2 prior lines of therapy for NSCLC, including participants with BRAF molecular alternations.
* Invasive malignancy or history of invasive malignancy other than disease under study within the last 2 years, except

  * Any other invasive malignancy for which the participant was definitively treated, has been disease-free for at least 2 years and in the opinion of the principal investigator and GlaxoSmithKline Medical Monitor will not affect the evaluation of the effects of the study treatment on the currently targeted malignancy, may be included in this clinical trial.
  * Curatively treated non-melanoma skin cancer or successfully treated in situ carcinoma.
* Carcinomatous meningitis (regardless of clinical status) and uncontrolled or symptomatic Central nervous system (CNS) metastases.
* Major surgery less than or equal to (<=) 28 days of first dose of study treatment.
* Autoimmune disease (current or history) or syndrome that required systemic treatment within the past 2 years. Replacement therapies which include physiological doses of corticosteroids for treatment of endocrinopathies (for example, adrenal insufficiency) are not considered systemic treatments.
* Receiving systemic steroids (>10 milligrams [mg]) oral prednisone or equivalent) or other immunosuppressive agents within 7 days prior to first dose of study treatment.
* Prior allogeneic/autologous bone marrow or solid organ transplantation.
* Receipt of any live vaccine within 30 days prior to first dose of study treatment.
* Toxicity from previous anticancer treatment that includes:

  1. Greater than or equal to (>=) Grade 3 toxicity considered related to prior immunotherapy and that led to treatment discontinuation.
  2. Toxicity related to prior treatment that has not resolved to <= Grade 1 (except alopecia, hearing loss, endocrinopathy managed with replacement therapy, and peripheral neuropathy which must be <= Grade 2).
* History (current and past) of idiopathic pulmonary fibrosis, pneumonitis (for past- pneumonitis exclusion only if steroids were required for treatment), interstitial lung disease, or organizing pneumonia.
* Recent history (within the past 6 months) of uncontrolled symptomatic ascites, pleural or pericardial effusions.
* Recent history (within the past 6 months) of gastrointestinal obstruction that required surgery, acute diverticulitis, inflammatory bowel disease, or intra-abdominal abscess.
* History or evidence of cardiac abnormalities within the 6 months prior to enrollment which include

  1. Serious, uncontrolled cardiac arrhythmia or clinically significant electrocardiogram abnormalities including second degree (Type II) or third degree atrioventricular block.
  2. Cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting or bypass grafting.
  3. Symptomatic pericarditis.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypo-albuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Active infection requiring systemic therapy <=7 days prior to first dose of study treatment.
* Participants with known human immunodeficiency virus infection.
* Participants with history of severe hypersensitivity to mAb or hypersensitivity to any of the study treatment(s) or their excipients.
* Participants requiring ongoing therapy with a medication that is a strong inhibitor or inducer of the cytochrome P 3A4 (CYP3A4) enzymes.
* Any serious and/or unstable pre-existing medical (aside from malignancy), psychiatric disorder, or other condition that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures in the opinion of the investigator.
* Pregnant or lactating female participants.
* Participant who is currently participating in or has participated in a study of an investigational device within 4 weeks prior to the first dose of study treatment.
* Participants with presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention.
* Participants with positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Participants with positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* Receipt of transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor, and recombinant erythropoietin) within 14 days before the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- GSK Investigational Site, Nashville, Tennessee, United States
- GSK Investigational Site, Brampton, Ontario, Canada
- GSK Investigational Site, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a sub-study of the master study NCT03739710. This sub study was terminated due to low enrolment of participants. The study was planned to include two phases - Part 1 and Part 2. No participants from this sub study were enrolled in part 2 as study was early terminated.
Groups:
- Feladilimab + Ipilimumab: Participants with Non-Small Cell Lung Cancer (NSCLC) received 24 milligram (mg) Feladilimab first as a 30-minute intravenous (IV) infusion followed by 1 mg/ kilogram (kg) Ipilimumab as IV infusion (started at least 30 minutes following the end of the feladilimab) once every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | Feladilimab + Ipilimumab
Started | 8
Completed | 0
Not Completed | 8
Not completed — Study Terminated by sponsor | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 8
Age, Customized [Number; unit: Participants]
  18 to 84 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race/Ethnicity, Customized [Number; unit: Participants] — Race categories (White and Asian where 0<n<11) are combined into 'All other races' category to maintain participant confidentiality and privacy.
  Participants
    All other races | 8

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or is a congenital anomaly/birth defect, other situations which involved medical or scientific judgment or is associated with liver injury and impaired liver function. SAEs are subset of AEs. AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA dictionary).
Time Frame: Up to 29 weeks
Population: Safety Population included all participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 8
Participants
  Any AE | 8
  Any SAE | 3

2. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Criteria for dose-limiting toxicity (DLT) included hematologic indicators such as febrile neutropenia as defined by CTCAE v5; Grade 4 neutropenia of >7 days in duration; Grade 4 anemia and Grade 3-4 thrombocytopenia with bleeding. Non-hematologic criteria, comprising Grade 4 toxicity; Grade 3 pneumonitis of any duration; Grade 3 toxicity that does not resolve to ≤Grade 1 or baseline within 3 days despite optimal supportive care; any Grade 2 ocular toxicity requiring systemic steroids, or any ≥ Grade 3 ocular toxicity Any other toxicity considered to be dose-limiting that occurs beyond four weeks was considered as DLT. Any other event which in the judgment of the investigator and GSK Medical Monitor is considered to be a DLT.
Time Frame: Up to 21 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 8
Participants | 2

3. Primary Outcome: Part 1: Number of Participants With Worst-case Change Post-baseline in Hematology Parameters
Description: Blood samples were collected for evaluation of hematology parameters. The summaries of worst-case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with decreases to low from baseline, changes to normal or no changes from baseline, and increases to high values have been presented. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Baseline (Day 1) and up to 29 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 8
Participants
  Basophils, Decrease to Low | 0
  Basophils, Change to Normal or No Change | 8
  Basophils, Increase to High | 0
  Eosinophils, Decrease to Low | 0
  Eosinophils, Change to Normal or No Change | 7
  Eosinophils, Increase to High | 1
  Erythrocytes, Decrease to Low | 2
  Erythrocytes, Change to Normal or No Change | 6
  Erythrocytes, Increase to High | 0
  Hemoglobin, Decrease to Low | 0
  Hemoglobin, Change to Normal or No Change | 8
  Hemoglobin, Increase to High | 0
  Ery. Mean Corpuscular HGB Concentration (EMCHC), Decrease to Low | 1
  EMCHC, Change to Normal or No Change | 7
  EMCHC, Increase to High | 0
  Ery. Mean Corpuscular Hemoglobin (EMCH), Decrease to Low | 0
  EMCH, Change to Normal or No Change | 7
  EMCH, Increase to High | 1
  Ery. Mean Corpuscular Volume (EMCV), Decrease to Low | 0
  EMCV, Change to Normal or No Change | 7
  EMCV, Increase to High | 1
  Hematocrit, Decrease to Low | 0
  Hematocrit, Change to Normal or No Change | 8
  Hematocrit, Increase to High | 0
  Leukocytes, Decrease to Low | 0
  Leukocytes, Change to Normal or No Change | 7
  Leukocytes, Increase to High | 1
  Lymphocytes, Decrease to Low | 0
  Lymphocytes, Change to Normal or No Change | 8
  Lymphocytes, Increase to High | 0
  Monocytes, Decrease to Low | 0
  Monocytes, Change to Normal or No Change | 7
  Monocytes, Increase to High | 1
  Neutrophils, Decrease to Low | 0
  Neutrophils, Change to Normal or No Change | 6
  Neutrophils, Increase to High | 2
  Platelets, Decrease to Low | 1
  Platelets, Change to Normal or No Change | 6
  Platelets, Increase to High | 1

4. Primary Outcome: Part 1: Number of Participants With Worst-case Change Post-baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for evaluation of clinical chemistry parameters. The summaries of worst-case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The number of participants with decreases to low from baseline, changes to normal or no changes from baseline, and increases to high values have been presented. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Baseline (Day 1) and up to 29 weeks
Population: Safety Population. Only those participants with data available in specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 8
Participants
  Alanine aminotransferase (ALT), Decrease to Low | 0
  ALT, Change to Normal or No Change | 6
  ALT, Increase to High | 2
  Albumin, Decrease to Low | 2
  Albumin, Change to Normal or No Change | 6
  Albumin, Increase to High | 0
  Alkaline Phosphatase (AP), Decrease to Low | 0
  AP, Change to Normal or No Change | 8
  AP, Increase to High | 0
  Aspartate Aminotransferase (AST), Decrease to Low | 0
  AST, Change to Normal or No Change | 8
  AST, Increase to High | 0
  Bilirubin, Decrease to Low | 0
  Bilirubin, Change to Normal or No Change | 8
  Bilirubin, Increase to High | 0
  C Reactive Protein (mg/L), Decrease to Low: number analyzed (Participants) | 3
  C Reactive Protein (mg/L), Decrease to Low | 0
  C Reactive Protein, Change to Normal or No Change: number analyzed (Participants) | 3
  C Reactive Protein, Change to Normal or No Change | 3
  C Reactive Protein, Increase to High: number analyzed (Participants) | 3
  C Reactive Protein, Increase to High | 0
  Calcium, Decrease to Low | 0
  Calcium, Change to Normal or No Change | 7
  Calcium, Increase to High | 1
  Creatinine, Decrease to Low | 1
  Creatinine, Change to Normal or No Change | 6
  Creatinine, Increase to High | 1
  Glucose, Decrease to Low | 0
  Glucose, Change to Normal or No Change | 7
  Glucose, Increase to High | 1
  Lactate Dehydrogenase (LDH), Decrease to Low | 0
  LDH, Change to Normal or No Change | 8
  LDH, Increase to High | 0
  Potassium, Decrease to Low | 1
  Potassium, Change to Normal or No Change | 7
  Potassium, Increase to High | 0
  Protein, Decrease to Low | 1
  Protein, Change to Normal or No Change | 7
  Protein, Increase to High | 0
  Sodium, Decrease to Low | 1
  Sodium, Change to Normal or No Change | 7
  Sodium, Increase to High | 0
  Thyrotropin, Decrease to Low: number analyzed (Participants) | 7
  Thyrotropin, Decrease to Low | 0
  Thyrotropin, Change to Normal or No Change: number analyzed (Participants) | 7
  Thyrotropin, Change to Normal or No Change | 5
  Thyrotropin, Increase to High: number analyzed (Participants) | 7
  Thyrotropin, Increase to High | 2
  Triiodothyronine, Free, Decrease to Low: number analyzed (Participants) | 4
  Triiodothyronine, Free, Decrease to Low | 1
  Triiodothyronine, Free, Change to Normal or No Change: number analyzed (Participants) | 4
  Triiodothyronine, Free, Change to Normal or No Change | 3
  Triiodothyronine, Free, Increase to High: number analyzed (Participants) | 4
  Triiodothyronine, Free, Increase to High | 0
  Troponin T, Decrease to Low: number analyzed (Participants) | 3
  Troponin T, Decrease to Low | 0
  Troponin T, Change to Normal or No Change: number analyzed (Participants) | 3
  Troponin T, Change to Normal or No Change | 2
  Troponin T, Increase to High: number analyzed (Participants) | 3
  Troponin T, Increase to High | 1
  Urea, Decrease to Low | 0
  Urea, Change to Normal or No Change | 3
  Urea, Increase to High | 5

5. Primary Outcome: Part 1: Number of Participants With Worst Case Change Post-baseline in Urinalysis Parameters
Description: Urine samples were collected for evaluation of urinalysis parameters using dipstick method. The dipstick test gave results in a semi-quantitative manner. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. The summaries of worst-case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with 'Any increase', or 'no changes/decreased' values have been presented.
Time Frame: Baseline (Day 1) and up to 29 weeks
Population: Safety Population. Only those participants with data available in specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 6
Participants
  Occult Blood, No Change/Decreased | 6
  Protein, Any Increase | 3
  Protein, No Change/Decreased | 3

6. Primary Outcome: Part 1: Change From Baseline in Potential of Hydrogen (pH) of Urine
Description: Urine samples were collected from participants to assess urine pH levels. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Changes from baseline in urine pH were reported.
Time Frame: Baseline (Day 1), week 4, week 7, week 10, week 13 and week 29 (Treatment Discontinuation)
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Potential of Hydrogen (pH)
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 6
Potential of Hydrogen (pH)
  Baseline (Day 1) | 6.33 (0.816)
  WEEK 4: number analyzed (Participants) | 5
  WEEK 4 | -0.80 (0.975)
  WEEK 7: number analyzed (Participants) | 2
  WEEK 7 | -0.50 (0.707)
  WEEK 10: number analyzed (Participants) | 1
  WEEK 10 | 0.00 (NA) — Standard deviation was not estimable for single participant.
  WEEK 13: number analyzed (Participants) | 1
  WEEK 13 | 0.50 (NA) — Standard deviation was not estimable for single participant.
  WEEK 29 (Treatment Discontinuation): number analyzed (Participants) | 3
  WEEK 29 (Treatment Discontinuation) | -0.50 (0.866)

7. Primary Outcome: Part 1: Change From Baseline in Specific Gravity of Urine
Description: Urine samples were collected from participants to analyze urine specific gravity. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Changes from baseline in specific gravity of urine were reported.
Time Frame: Baseline (Day 1), week 4, week 7, week 10, week 13 and week 29 (Treatment Discontinuation)
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Kilogram per cubic meter
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 6
Kilogram per cubic meter
  Baseline (Day 1) | 1.0175 (0.00418)
  WEEK 4: number analyzed (Participants) | 5
  WEEK 4 | 0.0050 (0.01173)
  WEEK 7: number analyzed (Participants) | 2
  WEEK 7 | 0.0150 (0.01414)
  WEEK 10: number analyzed (Participants) | 1
  WEEK 10 | 0.0000 (NA) — Standard deviation was not estimable for single participant
  WEEK 13: number analyzed (Participants) | 1
  WEEK 13 | 0.0250 (NA) — Standard deviation was not estimable for single participant.
  WEEK 29 (Treatment Discontinuation): number analyzed (Participants) | 3
  WEEK 29 (Treatment Discontinuation) | 0.0017 (0.00764)

8. Primary Outcome: Part 1: Number of Participants With AE Leading to Dose Modifications
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. The number of participants who experienced AE leading to dose modifications were evaluated.
Time Frame: Up to 29 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 8
Participants | 1

9. Primary Outcome: Part 2: Overall Survival
Description: OS is defined as the time from randomization until death due to any cause.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Part 1: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a confirmed complete response (CR) or confirmed partial response (PR) as their best overall response (BOR) recorded from the date of randomization until disease progression or initiation of new anti-cancer therapy, whichever is earlier based on blinded independent central review (BICR) evaluation criteria in solid tumors (RECIST) version 1.1 (v1.1). CR was defined as disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeter in the short axis. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters (e.g., percent change from baseline).
Time Frame: Up to 29 weeks
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 8
Percentage of participants
  Complete response | 0 [0 to 0]
  Partial response | 0 [0 to 0]

11. Secondary Outcome: Part 1: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a confirmed CR + PR at any time, plus stable disease (SD) >=12 weeks. PR was defined as at least 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm. Stable Disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: Up to 29 weeks
Population: Safety population. No participants had CR, PR, and SD.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

12. Secondary Outcome: Part 1: Maximum Concentration (Cmax) and Minimum Concentration (Cmin)
Description: Blood samples were collected for PK analysis.
Time Frame: Up to 29 weeks
Population: PK Population included all participants from the ITT Population from whom a blood sample is obtained and analyzed for PK concentration. As a result of the study termination, none of the participants had sufficient samples for analysis. Consequently, data was neither collected nor analyzed, and data will never be analyzed for this outcome measure in the future.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

13. Secondary Outcome: Part 2: Milestone Survival Rate at 12 and 18 Months
Description: Milestone survival rate is the proportion of participants who are alive at a specific, predefined point in time after a certain event or diagnosis post treatment.
Time Frame: At 12 and 18 months
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

14. Secondary Outcome: Part 2: Number of Participants With Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD) Based on RECIST 1.1
Description: Complete Response [CR], Partial Response [PR], stable disease [SD], and progressive disease (PD) as assessed by the investigator per IMWG. CR defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm; PR was defined as at least 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; Stable Disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

15. Secondary Outcome: Part 2: Number of Participants With iRECIST Complete Response (iCR), iRECIST Partial Response (iPR), iRECIST Stable Disease (iSD), iRECIST Confirmed Progressive Disease (iCPD), and iRECIST Unconfirmed Progressive Disease (iUPD)
Description: Modified RECIST 1.1 for immune-based therapeutics (iRECIST) is based on RECIST v 1.1 but adapted to account for the unique tumor response seen with immunotherapeutic drugs. iRECIST was to be used to assess tumor response and progression and make treatment decisions. iCR: disappearance of all target lesions; iPR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline). iCPD: either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; iSD: stable disease in the absence of CR or PD and iUPD: unconfirmed progressive disease when PD is unconfirmed.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

16. Secondary Outcome: Part 2: Number of Participants With PFS, ORR, DOR, and DCR
Description: PFS defined as time from the date of randomization to the date of disease progression or death, whichever will occurs earlier, per RECIST criteria. ORR defined as the percentage of participants with a confirmed CR or PR at any time per RECIST criteria. DOR defined as the time from first documented evidence of CR or PR until disease progression or death, per RECIST criteria. DCR was defined as the percentage of participants with a confirmed CR + PR at any time, plus stable disease (SD) >=12 weeks.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

17. Secondary Outcome: Part 2: Number of Participants With iPFS, iORR, and iDOR
Description: iPFS defined as time from the date of randomization to the date of disease progression or death, whichever will occurs earlier, per iRECIST criteria. iORR defined as the percentage of participants with a confirmed iCR or iPR at any time per iRECIST criteria. iDOR defined as the time from first documented evidence of CR or PR until disease progression or death, per iRECIST criteria.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

18. Secondary Outcome: Part 2: Number of Participants With AEs and SAEs
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function. AEs and SAEs were planned to be coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding system.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

19. Secondary Outcome: Part 2: Number of Participants With AESI
Description: Number of participants with AESI were planned to be evaluated.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

20. Secondary Outcome: Part 2: Number of Participants With AEs and SAEs Leading to Dose Modification
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function. AEs and SAEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding system. Number of participants with AEs and SAEs leading to dose modification (delays/withdrawal) were planned to be evaluated.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

21. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Changes in Hematology Lab Parameters
Description: Blood samples were to be collected for the analysis of hematology parameters. The laboratory parameters were to be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5. Grade 1 (G1): mild; Grade 2 (G2): moderate; Grade 3 (G3): severe or medically significant. Higher grade indicates greater severity and an increase in CTCAE grade were to be defined relative to the Baseline grade.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

22. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Changes in Clinical Chemistry Lab Parameters
Description: Blood samples were to be collected for the analysis of chemistry parameters. The laboratory parameters were to be graded according to CTCAE version 5. G1: mild; G2: moderate; G3: severe or medically significant. Higher grade indicates greater severity and an increase in CTCAE grade were to be defined relative to the Baseline grade.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

23. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs were planned to be measured after 5 minutes of rest and taken in the same position throughout the study.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

24. Secondary Outcome: Part 2: Maximum Concentration (Cmax) and Minimum Concentration (Cmin)
Description: Blood samples were planned to be collected for PK analysis.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

25. Secondary Outcome: Part 2: Number of Participants With Post-baseline Positive Anti-drug Antibodies (ADAs) Against Feladilimab
Description: Serum samples were to be collected for the analysis of the presence of ADAs using validated immunoassays.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

26. Secondary Outcome: Part 2: Number of Participants With Post-baseline Positive Anti-drug Antibodies (ADAs) Against Iplimumab
Description: Serum samples were to be collected for the analysis of the presence of ADAs using validated immunoassays.
Time Frame: Up to 29 weeks
Population: No participants were enrolled in Part 2 as study was terminated.
Arm/Group | Feladilimab + Ipilimumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to 29 weeks.
Description: Safety Population included all participants who received at least one dose of treatment.
Arm/Group | Feladilimab + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 4/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Feladilimab + Ipilimumab (N=8)
Pyrexia (General disorders) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Subacute inflammatory demyelinating polyneuropathy (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Feladilimab + Ipilimumab (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
General physical health deterioration (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebellar ataxia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Psychomotor retardation (Psychiatric disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT06790303/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT06790303/SAP_002.pdf